CLINICAL TRIAL: NCT01589328
Title: Randomized Controlled Trials for the Effect of Early Management on PAin and DEpression in Patients With PancreatoBiliary Cancer, EPADE-PB
Brief Title: Effect of Early Management on PAin and DEpression in Patients With PancreatoBiliary Cancer, EPADE-PB
Acronym: EPADE-PB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Sang Myung Woo, Staff physician, Ceneter for Liver Cancer, National Cancer Center, Korea
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NCCCTS-12-605
Record Dates: First submitted 2012-04-25; First posted 2012-05-01 (Estimated); Last update posted 2018-01-03 (Actual); Status verified 2018-01

CONDITIONS: Pancreatic Cancer; Biliary Tract Cancer; Cancer Pain; Depression
Keywords: pancreatic cancer; biliary tract cancer; cancer pain; depression
MeSH Terms: conditions — Pancreatic Neoplasms; Biliary Tract Neoplasms; Cancer Pain; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early Palliative care (Experimental): The interventions consisted of the following:
  (1) Nursing assessment of pain and depression mood (2) Pain control based NCCN guideline (3) Depression control by psychoeducation and/or consultation of psychiatrist specialist (4) Patient education
  Interventions: Other: Early Palliative care integrated with usual oncologic care
- Contol: usual oncologic care (No Intervention): Patients randomly assigned to usual oncologic care were not scheduled to meet with the palliative care service unless a meeting was requested by the patient, the family, or the oncologist; those who were referred to the service did not cross over to the early palliative care group or follow the specified palliative care protocol.

INTERVENTIONS:
Other: Early Palliative care integrated with usual oncologic care — Drug: The interventions consisted of the following:
  (1) Nursing assessment of pain and depression mood (2) Pain control based NCCN guideline (3) Depression control by psychoeducation and/or consultation of psychiatrist specialist (4) Patient education
  Other Names: Contol: usual oncologic care :NONE
  Arms: Early Palliative care

SUMMARY:
Effect of Early management on PAin and DEpression in patients with PancreatoBiliary Cancer, EPADE-PB

Purpose

To determine whether early palliative care integrated with usual oncologic care with automated symptom monitoring can improve depression and pain in patients with cancer

ELIGIBILITY:
Inclusion Criteria:

* Ages Eligible for Study: 18 Years and older Genders Eligible for Study: Both Accepts Healthy Volunteers: No
* Pathologic confirmed locally advanced or metastatic pancreatic cancer or biliary tract cancer
* within 8 weeks after diagnosis
* cancer-related pain (Brief Pain Inventory [BPI] worst pain score >3), depression (Center for Epidemiological Studies-Depression Scale [CES-D] >16) or both
* Karnofsky Performance Rating Scale ≥50%

Exclusion Criteria:

* Opioid intolerance
* History of drug or alcohol abuse
* Impaired sensory or cognitive function
* Pregnant or lactating woman
* Women of child bearing potential not using a contraceptive method
* Sexually active fertile men not using effective birth control during medication of study drug and up to 6 months after completion of study drug if their partners are women of child-bearing potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2012-03-15 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Reduction in pain score | at baseline, 1 month, and every 3 months, up to 1 year
  • Reduction in pain scores, Brief Pain Inventory [BPI] severity
Reduction in depression score | at baseline, 1 month, and every 3 months, up to 1 year
  Reduction in depression score, Center for Epidemiological Studies-Depression Scale [CES-D]

SECONDARY OUTCOMES:
Quality of life | at baseline, 1 month, and every 3 months, up to 1 year
  EORTC QLQ-C30 General Questionnaire, Korean version
Overall survival | at baseline, 1 month, and every 3 months, up to 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center, Goyang, 410-769, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No